CLINICAL TRIAL: NCT00416364
Title: The Economic Impact of Four Varieties of Mesh Inguinal Hernia Repair- a Double-Blinded, Prospective, Randomized Trial
Status: Terminated | Type: Observational
Why Stopped: Inadequate accrural rates
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: CAPT Paul Lucha, NMCP
Other Study IDs: P06-020
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Inguinal Hernia
Keywords: hernia; inguinal; quality of life
MeSH Terms: conditions — Hernia, Inguinal; Hernia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1
- 2
- 3
- 4

SUMMARY:
There are a variety of methods to repair inguinal hernias. Each has its advocate and may confer advantages to individual patients. Postoperative pain, convalescence, recurrence, and economics have all been evaluated however none in a randomized blinded fashion. Recently, investigators have attempted to address some of these concerns with new prosthetic materials. The preferred method of repair currently employs a tension free technique using mesh prosthesis. The approach as advocated by Lichtenstein involves reinforcing the floor of the inquinal canal with an onlay mesh. Newer approaches use a double layer mesh that reinforces the floor in a preperitoneal and onlay technique (Prolene Hernia System) while obliterating the internal inguinal ring or by the Mesh Plug repair (bioresorbable or permanent) which reinforces the inguinal floor with an onlay mesh while obliterating the internal inguinal ring. Currently no study has compared these techniques for ease of performance, postoperative pain, convalescence, quality of life, or cost in a randomized double blinded fashion. NMCP is uniquely qualified to compare these repairs prospectively and blinded to best assess the most cost effective approach which causes the least pain. A prospective double-blinded randomized trial comparing the Lichtenstein onlay mesh technique to Prolene Hernia Sytem (PHS), Mesh Plug Repair (MPR), or Gore Bioresorbable plug for postoperative pain, duration of convalescence, cost, impact on quality of life and ease of performance is proposed. Impact on quality of life will be assessed serially with the SF 12 which is a validated survey used with serial measures in the acute setting.

DETAILED DESCRIPTION:
4. RESEARCH DESIGN/METHODS/SUBJECT JUSTIFICATION

1. General Approach To randomize between Lichtenstein, PHS, GBP,and MPR hernia repair in a double blinded fashion in patients presenting to the general surgery clinic with primary unilateral inguinal hernias. . Daily visual analogue pain scales (validated for this purpose) will be obtained. An SF 12, quality of life instrument, validated for this purpose will be provided on a weekly basis to assess impact, if any, that differing hernia repairs may have. This instrument has been validated to provide serial assessments in quality of life in surgical patients.

   (1) Research Objective 2. Comparison of operative costs between groups. 3. Comparison of Visual Analogue Pain Scale between groups to assess differences in percieved postoperative pain.

   4. Comparison of operative times between groups as an estimation of operative ease in performing the different procedures.

   5. Comparison of Quality of life suveys (SF 12) serially between groups.

   (2) Detail how many groups or arms are in the study and what each receives Patients will be assigned randomly to one of four comonly performed hernia repairs; Lichtenstein, MPR, GBP, and PHS. See below for details in the procedures.

   (3) Randomization Procedures Computer generated block randomized list will assign patients to one of four repairs on the morning of surgery.
2. Methods and Materials

   1. Lichtenstein hernia repair: A piece of polyproplene mesh will be trimmed to fit the inguinal floor. The mesh will be secured to poupart's ligament and the conjoined tendon using 2-0 prolene suture. Tacking sutures of 2-0 Vicryl will be used laterally to secure the mesh in place.
   2. Mesh Plug hernia repair (MPR): A 2 part prosthesis (Perfix Plug) is fixed in place using 2-0 vicryl. The plug is secured into the inguinal ring and the onlay mesh is tacked to the same structures noted for the Lichtenstein hernia repair using 2-0 Vicyrl.
   3. Prolene Hernia System (PHS): The preperitoneal space is developed through the internal ring. The inner mesh is placed beneath the transversalis fascia and the superficial mesh sits above the transversalis fascia. The outer mesh is fixed with tacking sutures to the same structures noted for the Lichtenstein hernia repair using 2-0 Vicyrl.
   4. Gore Bioresorbable Plug (GBP): The plug is secured to the internal inguinal ring with 2-0 Vicryl.

Closure of the fascia of the external oblique, scarpa's fascia and skin will be accomplished with 2-0 vicryl (fascia) and 4-0 monocryl sutures for all hernia repairs. Postoperative management of pain will include oral narcotics and non steroidal anti inflammaory medication.

The active duty male patients with primary unilaterial inguinal hernia seen in the General Surgery Clinic will be offered participation in the protocol. An investigator or Subinvestigator will explain the details of the study to eligible patients and if interested, they will consent said patients. They will be randomized the morning of the operative procedure. On discharge, the surgeon will recommend convalescent leave based on their individual preferances (this is current standard of care) and the patient will be asked to record their visual analogue pain scales daily. They will be seen in the surgery clinic before expiration of the con leave and re assessed for additional need for con leave by a clinic nurse (unaware of which surgical procedure the patient had ) who will provide recommendations for additional con leave to the responsible surgeon. The patient will be contacted weekly by and investigator and the telephone version of the SF12 will be administered until 30 days postoperatively (4 samples). The responsible surgeon has final responsibility for recommendation of con leave. . Operative times will be recorded from the operative record and costs will be generated from actual material costs and an average of OR room charges and anesthesia charges from the tidewater area.

1. Standard of Care Primary inguinal hernias are repaired in a tension free fashion. The lichtenstein, mesh plug repair, bioresorbable plug, and prolene hernia system are commonly performed repairs. Surgeons choose one of these repairs based on personal preference and ease of performance.
2. Experimental Procedure Randomization and blinding between hernia repair types, collecting pain data (VAS), costs, and quality of life questionaires.

We have propose the following changes to the protocol which have been submitted to the IRB to facilitate enrollment. The protocol was approved in February 2006 with an anticipated enrollment requirement of 680 patients. To date, one patient has enrolled. The majority of patients have declined participation because they prefer not to return to the clinic weekly until returning to work. As return to work and con leave were not primary end points of the study (operative times, VAS, and QOL are the endpoints of interest), the following changes are recommended to improve participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral primary inguinal hernia presenting for repair

Exclusion Criteria:

* Recurrent repairs
* Females
* Bilateral repairs
* Repairs done with other operative procedures

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AD males with primary hernia
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2006-03; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Comparison of Visual Analogue Pain Scale between groups to assess differences in percieved postoperative pain. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Lucha, DO, Principal Investigator — Naval Medical Center Department of Surgery- Portsmouth, VA
Locations (1):
- Naval Medical Center Department of Surgery, Portsmouth, Virginia, United States